CLINICAL TRIAL: NCT00805831
Title: Safety and Efficacy of Using HDH Device and Method - a Novel Sutureless Vascular Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HDH Medical Ltd (Industry)
Responsible Party: Dr. Hanna Levy, Clinical Study Consultant, Qsite
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDH -AAA-P-01
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Vascular Disease; Atherosclerosis
Keywords: sutureless vascular bypass
MeSH Terms: conditions — Vascular Diseases; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Aortic anastomosis surgery will be conducted using HDH device.
  Interventions: Device: HDH

INTERVENTIONS:
Device: HDH — sutureless vascular anastomosis

SUMMARY:
The HDH device is intended for creating sutureless vascular anastomosis in various blood vessels. The HDH device consists of four parts: an elastic tube (graft), docking head (anastomotic device), inversion device (connects the vascular graft to HDH) and measuring device. This study was design in order to evaluate the safety and efficacy of using HDH device and method an innovative anastomotic device for sutureless aortic anastomosis in patient diagnosed with abdominal aneurysm or Aorto-iliac aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Patient age above 18 (men and woman)
* Patient suffers from infrarenal abdominal aortic or Aorto-iliac aneurysm
* Aneurysm diameter is larger than 5cm/ its annual growth is more than 0.5cm/or iliac aneurysm size is larger than 2.5cm
* The abdominal aneurysm neck is longer than 1.5 cm
* Patient's physical condition allows performing general anesthesia
* Patient is willing to sign the informed consent and follow the study protocol.

Exclusion Criteria:

* Patient Age under 18 years
* Patient's physical condition dose not allows to perform general anesthesia
* Patient's with terminal disease and life expectancy of less than 3 months
* Patient objects to the treatment or study protocol
* Anesthesiologist or personal care physician object
* Patient suffer from Supra/infrarenal AAA
* The abdominal aneurysm neck is smaller than 1.5 cm
* Aneurysm diameter is smaller than 5cm/ its annual growth is less than 0.5cm/

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To establish safety of using the HDH device for creating sutureless aortic anastomosis. Safety will be established by lack of serious adverse events. | within 1 month

SECONDARY OUTCOMES:
Time to complete the anastomosis | during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Boris Yofee, MD, Principal Investigator — Barzilai Medical Center, Ashkelon, Israel
Locations (1):
- Barzilai Medical center, Ashkelon, Israel